CLINICAL TRIAL: NCT05929703
Title: Evaluating Novel Healthcare Approaches to Nurturing and Caring for Hospitalized Elders (ENHANCE)
Brief Title: Evaluating Novel Healthcare Approaches to Nurturing and Caring for Hospitalized Elders
Acronym: ENHANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Hebrew SeniorLife (Other); MaineHealth (Other); University of Pennsylvania (Other); West Penn Allegheny Health System (Other); UnityPoint Health - Meriter Hospital (Unknown); University of Utah (Other); MemorialCare Saddleback Medical Center (Unknown); Brandeis University (Other); Indiana University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Phillip Vlisides, Assistant Professor of Anesthesiology; Executive Director, Neuroscience Research, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HUM00227397; DE-2022C1-25666 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2023-06-20; First posted 2023-07-03 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Delirium; Neurocognitive Disorders; Mild Cognitive Impairment; Alzheimer Disease; Aging; Family Support; Family Members; Caregiver Burden; Implementation Science; Patient Satisfaction
Keywords: Delirium; Clinical Trial; Comparative Effectiveness Research; Implementation Science
MeSH Terms: conditions — Delirium; Neurocognitive Disorders; Cognitive Dysfunction; Alzheimer Disease; Caregiver Burden; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Stepped-wedge, cluster randomized
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hospital Elder Life Program (HELP) (Active Comparator): Hospital Elder Life Program (HELP) is built upon multicomponent, non-pharmacologic strategies that target delirium risk factors to optimize cognitive and clinical function during hospitalization.
  Interventions: Behavioral: HELP
- Family-Augmented Hospital Elder Life Program (FAM-HELP) (Active Comparator): The FAM-HELP program will incorporate a family member and/or care partner, who will play a central role with providing bedside support for delirium risk reduction. Family members and care partners will provide social and emotional support along with augmentation of HELP-based protocols.
  Interventions: Behavioral: FAM-HELP

INTERVENTIONS:
Behavioral: HELP — This is usual (standard) care across hospitals in this trial. A multidisciplinary team of nurse specialists, social workers, and volunteers implement daily protocols focused on orientation, cognitive stimulation, early mobilization, sleep enhancement, support with visual and hearing aids, mealtime assistance, hydration, reduction in polypharmacy, and nursing-based delirium prevention protocols.
  Arms: Hospital Elder Life Program (HELP)
Behavioral: FAM-HELP — Family members and care partners will provide daily emotional and social support during hospitalization. Additionally, family members and care partners will engage in HELP-based protocols throughout the day. The rationale for this protocol augmentation is two-fold: (1) HELP may not consistently have available volunteers (e.g., short-staffing) during a hospital stay, and (2) patients may be more likely to engage in therapeutic activities with a family member given the connection and comfort level.
  Arms: Family-Augmented Hospital Elder Life Program (FAM-HELP)

SUMMARY:
The goal of this clinical trial is to compare the Hospital Elder Life Program (HELP) with a family-augmented version of HELP (FAM-HELP), that includes family members and care partners, for the prevention of delirium in older patients during hospital admission. The main objectives of the trial are the following:

1. To compare the effectiveness of FAM-HELP and HELP in reducing both the incidence of delirium and its severity.
2. To compare the effectiveness of FAM-HELP and HELP in improving patient- and family-reported outcomes.
3. To explore the implementation context, process, and outcomes of the FAM-HELP program in diverse hospital settings.

DETAILED DESCRIPTION:
Delirium is a common complication of hospitalization and major surgery for older adults, and it can lead to loss of independence and substantial healthcare costs. One approach to preventing delirium is through the Hospital Elder Life Program (HELP). HELP personnel work to prevent delirium by providing orienting communication, assisting patients with walking and exercise, providing help with nutrition and fluids, implementing sleep protocols, and helping patients with vision and hearing aids.

However, it is unknown whether involving family members in these activities along with HELP staff (i.e., "FAM-HELP") might be more effective with preventing delirium. The objective of this clinical trial is thus to compare the traditional HELP program with a family-augmented version of HELP (FAM-HELP) to determine which program is more effective with preventing delirium and related complications in older, hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* At least 70 years of age
* Anticipated length of hospital stay at least 72 hours
* Family member or care partner available to be on-site in the hospital
* At least one delirium risk factor (e.g., cognitive or functional impairment, dehydration, vision or hearing impairment)
* Evaluable cognitive function at baseline (i.e., ability to complete baseline cognitive function assessment)

Exclusion Criteria:

* Delirium on admission
* Unable to communicate verbally (e.g., coma, mechanical ventilation)
* Unable to participate fully in interventions (e.g., terminal condition, advanced dementia)
* Staff safety concerns (e.g., violent behavior)
* Cardiac or intracranial surgery (due to competing causes of delirium)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Delirium Incidence | Day of trial enrollment through day of hospital discharge, up to 14 days
  Any positive delirium screen (yes/no) as determined by the long-form Confusion Assessment Method (CAM), supplemented by a validated chart review approach for delirium.
Delirium Severity | Day of trial enrollment through day of hospital discharge, up to 14 days
  Delirium severity will be scored using the Confusion Assessment Method Long Form Severity Score (CAM-S) (n, 0-19, with higher number indicating more severe delirium). Score derived from the same CAM instrument and items used for delirium incidence.

SECONDARY OUTCOMES:
Delirium Duration | Day of trial enrollment through day of hospital discharge, up to 14 days
  The cumulative number of days (n) with a positive delirium screen will be calculated for all participants
Persistent Delirium | 30 days after hospital discharge
  Positive delirium screen (yes/no) 30 days after hospital discharge as determined by the long-form Confusion Assessment Method (AM)
Delirium Burden - Patient | Day of trial enrollment through 30 days after discharge
  Delirium burden will be calculated using the Patient Delirium Burden Scale (DEL-B-P) (n, 0-40, with higher number indicating more severe burden)
Delirium Burden - Family and Care Partners | Day of trial enrollment through 30 days after discharge
  Delirium burden will be calculated using the Patient Delirium Family Caregiver Scale (DEL-B-C) (n, 0-40, with higher number indicating more severe burden)
Caregiving Strain | Hospital discharge through 30 days after discharge
  Strain associated with patient caregiving will be assessed via Modified Caregiver Strain Index (MCSI) (n, 0-26, with higher number indicating more caregiver strain)
Cognitive Function - Subjective Reporting | Hospital discharge through 30 days after discharge
  Subjective reporting of cognitive function will be assessed via PROMIS Cognitive Function - Short Form 6a (n, 6-30, with higher number indicating better subjective cognitive function)
Hospital Experience | Day of hospital discharge (typically up to 30 days after hospital admission, may extend to 60 or more days)
  Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) Survey (n, 7-28, with higher score indicating better hospital experience)
Global Health | Hospital discharge through 30 days after discharge
  Assessment of overall physical and mental health via PROMIS Global Health-10. Two separate subscales will be calculated, Global Physical Health (n, 4-20) and Global Mental Health (n, 4-20), with higher scores indicating better health.
Physical Function | 30 days after hospital discharge
  Assessment of physical function via PROMIS Physical Short Form 10a (n, 10-50, with higher scores indicating better physical function).
Falls | Day of trial enrollment through 30 days after hospital discharge
  Proportion of participants in each group (%) experiencing at least one fall
Length of Hospital Stay | Day of hospital admission through hospital discharge (typically up to 30 days after hospital admission, may extend to 60 or more days)
  Total number of days (n) spent in the hospital
Discharge Disposition | Day of hospital discharge through 30 days after discharge
  Proportion of patients in each group (%) discharged somewhere other than home (e.g., Long-Term Care Facility)
30-Day Readmission | Day of hospital discharge through 30 days after discharge
  Proportion of participants in each group (%) requiring hospital readmission

OTHER OUTCOMES:
Antipsychotic use | Day of trial enrollment through day of hospital discharge, up to 14 days
  Proportion of participants in each group (%) requiring antipsychotic medications during hospitalization
Restraint use | Day of trial enrollment through day of hospital discharge, up to 14 days
  Proportion of participants in each group (%) requiring restraint use during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Sharon K Inouye, MD, Principal Investigator — Hebrew SeniorLife; Phillip E Vlisides, MD, Principal Investigator — University of Michigan
Locations (7):
- United States (7):
  - Saddleback Medical Center, Orange, California
  - MaineHealth, Portland, Maine
  - Michigan Medicine, Ann Arbor, Michigan
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Meriter Hospital, Madison, Wisconsin